CLINICAL TRIAL: NCT00741169
Title: Phase I, Open-label, 3-way Crossover Trial in Healthy Volunteers to Determine the Drug-drug Interaction Between TMC435350 and Rifampin After Multiple Dosing.
Brief Title: TMC435350-TiDP16-C105: Phase I, 3-way Crossover, Drug-drug Interaction Between TMC435350 and Rifampin After Multiple Dosing.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015412
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C; HCV; Tuberculosis; Rifampin; Pharmacokinetics
Keywords: TMC435350-TiDP16-C105; TMC435350-C105; Hepatitis C; HCV; Rifampin
MeSH Terms: conditions — Hepatitis C; Tuberculosis | interventions — Simeprevir; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence will consist of Treatment A (TMC435350 200 mg once daily for 7 days), Treatment B (rifampin 600 mg once daily for 7 days), and Treatment C (TMC435350 200 mg once daily+rifampin 600 mg once daily for 7 days). Participants will receive 1 treatment (A, B, or C) during each treatment session. There will be 3 treatment sessions, each treatment session will be separated by 10 days.
  Interventions: Drug: TMC435350; Drug: Rifampin; Drug: TMC435350+rifampin
- Treatment Sequence BCA (Experimental)
  Interventions: Drug: TMC435350; Drug: Rifampin; Drug: TMC435350+rifampin
- Treatment Sequence CAB (Experimental)
  Interventions: Drug: TMC435350; Drug: Rifampin; Drug: TMC435350+rifampin
- Treatment sequence CBA (Experimental)
  Interventions: Drug: TMC435350; Drug: Rifampin; Drug: TMC435350+rifampin
- Treatment Sequence BAC (Experimental)
  Interventions: Drug: TMC435350; Drug: Rifampin; Drug: TMC435350+rifampin
- Treatment Sequence ACB (Experimental)
  Interventions: Drug: TMC435350; Drug: Rifampin; Drug: TMC435350+rifampin

INTERVENTIONS:
Drug: TMC435350 — 200 mg taken by mouth once daily for 7 days
Drug: Rifampin — 600 mg taken by mouth once daily for 7 days
Drug: TMC435350+rifampin — The combination of TMC435350 200 mg + rifampin 600 mg both taken by mouth once daily for 7 days.

SUMMARY:
The purpose of this study is to assess the interactions seen when somebody doses with TMC435350 and Rifampin (commercial form of antibiotic).

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized, 3-way crossover trial in 18 healthy volunteers to investigate the potential drug-drug interaction between rifampin and TMC435350. TMC435350 is a protease inhibitor in development for treatment of chronic HCV infection. The goal is to assess the PK and safety data generated during 3 in-patients sessions. At each session the volunteer will receive one of 3 treatments. Rifampin is a medication commonly given to patients with Mycobacterium infections such as tuberculosis. Some patients have both chronic HCV and tuberculosis, therefore it is necessary to know how the medications will affect each other when they are taken together. Treatment A: TMC435350 200 mg q.d. for 7 days. Treatment B: rifampin 600 mg q.d. for 7 days. Treatment C: the combination of TMC435350 200 mg q.d. + rifampin 600 mg q.d. for 7 days. There will be a washout period of at least 10 days between subsequent sessions. Day 8 of a treatment session is the first day of the washout period. Full pharmacokinetic profiles of TMC435350 will be determined on Day 7 of Treatments A and C. Full pharmacokinetic profiles of rifampin and its active metabolite 25-deacetyl rifampin will be determined on Day 7 of Treatments B and C. Safety and tolerability will be monitored continuously throughout the trial. Volunteers will receive the dose regimens in Treatments A, B, C: Treatment A: TMC435350 200 mg q.d. for 7 days. Treatment B: rifampin 600 mg q.d. for 7 days, Treatment C: the combination of TMC435350 200 mg+rifampin 600 mg both q.d. for 7 days. The volunteers will enter the testing facility the night before the first dosing in each session (on Day -1 = one day before the first dosing) and stay in the testing facility until 72 hours after the last intake of medication on Day (10).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet all of the following inclusion criteria: Non smoking for at least 3 months prior to selection, Normal weight as defined by a body mass index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 32.0 kg/m2, extremes included), Informed Consent Form (ICF) signed voluntarily before the first trial related activity, Able to comply with protocol requirements, Normal 12-lead electrocardiogram (ECG) (in triplicate) at screening including: Normal sinus rhythm (heart rate [HR] between 40 and 100 bpm), QTc interval = 450 ms, QRS interval < 120 ms, PR interval = 220 ms
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, vital signs, and the results of blood biochemistry, and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* Past history of heart arrhythmias (extrasystole, tachycardia at rest) or having baseline prolongation of QTc interval > 450 ms
* history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT syndrome)
* Female, except if postmenopausal since more than 2 years, or posthysterectomy, or post tubal ligation (without reversal operation)
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the trial procedures
* Hepatitis A, B, or C infection (confirmed by hepatitis A antibody, hepatitis B surface antigen, or hepatitis C virus antibody, respectively) or human immunodeficiency virus - type 1 (HIV-1) or HIV-2 infection at screening
* A positive urine drug test at screening
* Currently active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* Currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability
* Any history of significant skin disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of TMC435350 | On Day 1, 2, 4, 6, and 7 of Treatments A and C
  The following PK parameters will be assessed: C0h on Day 7 of Treatments A and C; and C0h, Cmin, Cmax, tmax, AUC24h, Css,av, FI, λz, t1/2term, Ratio Cmin test/ref, Ratio C0h test/ref, Ratio Cmax test/ref, and Ratio AUC24h test/ref.
Pharmacokinetic (PK) profile of rifampin and 25-deacetylrifampin | On Day 1, 2, 4, 6, and 7 of Treatments B and C
  The PK parameter of C0h will be assessed on Day 1, 2, 4 and 6 of Treatments B and C, and the PK parameters of C0h, Cmin, Cmax, tmax, AUC24h, Css,av, FI, λz, t1/2term, Ratio Cmin test/ref, Ratio C0h test/ref , Ratio Cmax test/ref , Ratio AUC24h test/ref on Day 7 of Treatments B and C.

SECONDARY OUTCOMES:
The number of participants reporting adverse events as a measure of safety and tolerability. | Up to 30 to 35 days after the last intake of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited